CLINICAL TRIAL: NCT02121847
Title: Investigation of Maintaining Visual Performance Achieved With Cyclosporine Therapy
Acronym: IMPACT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GMA-RES-014-001
Record Dates: First submitted 2014-04-22; First posted 2014-04-24 (Estimated); Results first posted 2016-04-25 (Estimated); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Dry Eye Syndromes
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Cyclosporine; Cyclosporins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- cyclosporine 0.05% ophthalmic emulsion (Experimental): Cyclosporine 0.05% ophthalmic emulsion (Restasis®) eye drops administered twice daily and carboxymethylcellulose-based lubricant eye drops (Refresh OPTIVE® Advanced) administered as needed for 6 months.
  Interventions: Drug: cyclosporine 0.05% ophthalmic emulsion; Drug: carboxymethylcellulose-based lubricant eye drops

INTERVENTIONS:
Drug: cyclosporine 0.05% ophthalmic emulsion — Cyclosporine 0.05% ophthalmic emulsion (Restasis®) eye drops administered twice daily for 6 months.
  Other Names: Restasis®
Drug: carboxymethylcellulose-based lubricant eye drops — Carboxymethylcellulose-based lubricant eye drops (Refresh OPTIVE® Advanced) administered as needed for 6 months.
  Other Names: Refresh OPTIVE® Advanced

SUMMARY:
This study will evaluate the safety and efficacy of cyclosporine 0.05% ophthalmic emulsion (Restasis®) in patients with dry eye disease.

ELIGIBILITY:
Inclusion Criteria:

* History of dry eye in both eyes
* Willing to use eye drops for dry eye symptoms

Exclusion Criteria:

* Anticipate wearing contact lenses during the study
* Laser-assisted in situ keratomileusis (LASIK) surgery within the past 12 months
* Any ocular and/or lid surgeries within the past 6 months
* Cataract surgery in either eye
* Current or anticipated use of temporary punctal plugs during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-04-03 (Actual); Primary Completion 2014-09-23 (Actual); Study Completion 2014-09-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- Andover, Massachusetts, United States

REFERENCES:
- [Background] Stonecipher KG, Torkildsen GL, Ousler GW 3rd, Morris S, Villanueva L, Hollander DA. The IMPACT study: a prospective evaluation of the effects of cyclosporine ophthalmic emulsion 0.05% on ocular surface staining and visual performance in patients with dry eye. Clin Ophthalmol. 2016 May 13;10:887-95. doi: 10.2147/OPTH.S101627. eCollection 2016. PMID 27257373

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cyclosporine 0.05% Ophthalmic Emulsion
Started | 40
Completed | 37
Not Completed | 3
Not completed — Administrative Reasons | 1
Not completed — Adverse Event | 2

BASELINE CHARACTERISTICS:
Arm/Group | Cyclosporine 0.05% Ophthalmic Emulsion
Number analyzed (Participants) | 40
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.4 (9.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35
  Male | 5

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Total Corneal Staining Score With Fluorescein in the Worse Eye
Description: Total corneal staining with fluorescein is measured in the worse eye utilizing the Ora CalibraTM Corneal Flourescein Staining Scale (0 to 4 scale where 0=no staining and 4= severe staining). The sum of the total includes 3 regions of the cornea, resulting in a maximum possible score of 12 (severe staining score of 4 in all three regions). A negative change from baseline represents a decrease in staining (improvement). A positive change from baseline represents an increase in staining (worsening).
Time Frame: Baseline, Month 6
Population: Intent-to-Treat: all enrolled patients who received at least one dose of the study drug
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Cyclosporine 0.05% Ophthalmic Emulsion
Number analyzed (Participants) | 40
Scores on a Scale
  Baseline | 7.29 (1.409)
  Change from Baseline at Month 6 (N=37) | -1.96 (1.677)

2. Primary Outcome: Change From Baseline in Total Conjunctival Staining Score With Fluorescein in the Worse Eye
Description: Total conjunctival staining with fluorescein is measured in the worse eye utilizing the Ora CalibraTM Conjunctiva Flourescein Staining Scale (0 to 4 scale where 0=no staining and 4= severe staining). The sum of the total includes 2 regions of the conjunctiva, resulting in a maximum possible score of 8 (severe staining score of 4 in both regions). A negative change from baseline represents a decrease in staining (improvement). A positive change from baseline represents an increase in staining (worsening).
Time Frame: Baseline, Month 6
Population: Intent-to-Treat: all enrolled patients who received at least one dose of the study drug
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Cyclosporine 0.05% Ophthalmic Emulsion
Number analyzed (Participants) | 40
Scores on a Scale
  Baseline | 4.68 (1.035)
  Change from Baseline at Month 6 (N=37) | 0.11 (1.162)

3. Primary Outcome: Change From Baseline in Total Corneal Staining Score With Lissamine Green in the Worse Eye
Description: Total corneal staining with lissamine green is measured in the worse eye utilizing the Ora CalibraTM Corneal Lissamine Staining Scale (0 to 4 scale where 0=no staining and 4= severe staining). The sum of the total includes 3 regions of the cornea, resulting in a maximum possible score of 12 (severe staining score of 4 in all three regions). A negative change from baseline represents a decrease in staining (improvement). A positive change from baseline represents an increase in staining (worsening).
Time Frame: Baseline, Month 6
Population: Intent-to-Treat: all enrolled patients who received at least one dose of the study drug
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Cyclosporine 0.05% Ophthalmic Emulsion
Number analyzed (Participants) | 40
Scores on a Scale
  Baseline | 4.43 (1.389)
  Change from Baseline at Month 6 (N=37) | -0.93 (1.439)

4. Primary Outcome: Change From Baseline in Total Conjunctival Staining Score With Lissamine Green in the Worse Eye
Description: Total conjunctival staining with lissamine is measured in the worse eye utilizing the Ora CalibraTM Conjunctiva Lissamine Staining Scale (0 to 4 scale where 0=no staining and 4= severe staining). The sum of the total includes 2 regions of the conjunctiva, resulting in a maximum possible score of 8 (severe staining score of 4 in both regions). A negative change from baseline represents a decrease in staining (improvement). A positive change from baseline represents an increase in staining (worsening).
Time Frame: Baseline, Month 6
Population: Intent-to-Treat: all enrolled patients who received at least one dose of the study drug
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Cyclosporine 0.05% Ophthalmic Emulsion
Number analyzed (Participants) | 40
Scores on a Scale
  Baseline | 4.21 (1.255)
  Change from Baseline at Month 6 (N=37) | 0.30 (1.356)

5. Primary Outcome: Change From Baseline in Reading on the Ocular Surface Disease Index (OSDI)
Description: The OSDI consists of 12 questions measuring the presence of ocular symptoms. The reading question is assessed using a 5-point scale (0=none of the time; 4=all of the time). The reading score is converted to a 0-100 score where 0 is best and 100 is worst. Higher OSDI reading scores are associated with greater severity. A negative number change from baseline indicates improvement and a positive number change from baseline indicates worsening.
Time Frame: Baseline, Month 6
Population: Intent-to-Treat: all enrolled patients who received at least one dose of the study drug
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Cyclosporine 0.05% Ophthalmic Emulsion
Number analyzed (Participants) | 40
Scores on a Scale
  Baseline | 1.4 (1.11)
  Change from Baseline at Month 6 (N=36) | -0.7 (1.07)

6. Primary Outcome: Change From Baseline in Driving at Night on the OSDI
Description: The OSDI consists of 12 questions measuring the presence of ocular symptoms. The driving at night question is assessed using a 5-point scale (0=none of the time; 4=all of the time). The driving at night score is converted to a 0-100 score where 0 is best and 100 is worst. Higher OSDI reading scores are associated with greater severity. A negative number change from baseline indicates improvement and a positive number change from baseline indicates worsening.
Time Frame: Baseline, Month 6
Population: Intent-to-Treat: all enrolled patients who received at least one dose of the study drug and who have data for this outcome measure
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Cyclosporine 0.05% Ophthalmic Emulsion
Number analyzed (Participants) | 35
Scores on a Scale
  Baseline | 2.3 (1.46)
  Change from Baseline at Month 6 (N=28) | -0.5 (1.32)

7. Primary Outcome: Change From Baseline in Working With a Computer or Bank Machine on the OSDI
Description: The OSDI consists of 12 questions measuring the presence of ocular symptoms. The working with a computer or bank machine question is assessed using a 5-point scale (0=none of the time; 4=all of the time). The working with a computer or bank machine score is converted to a 0-100 score where 0 is best and 100 is worst. Higher OSDI reading scores are associated with greater severity. A negative number change from baseline indicates improvement and a positive number change from baseline indicates worsening.
Time Frame: Baseline, Month 6
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Cyclosporine 0.05% Ophthalmic Emulsion
Number analyzed (Participants) | 38
Scores on a Scale
  Baseline | 2.2 (1.10)
  Change from Baseline at Month 6 (N=34) | -1.0 (1.06)

8. Primary Outcome: Change From Baseline in Watching TV on the OSDI
Description: The OSDI consists of 12 questions measuring the presence of ocular symptoms. The watching TV question is assessed using a 5-point scale (0=none of the time; 4=all of the time). The watching TV score is converted to a 0-100 score where 0 is best and 100 is worst. Higher OSDI reading scores are associated with greater severity. A negative number change from baseline indicates improvement and a positive number change from baseline indicates worsening.
Time Frame: Baseline, Month 6
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Cyclosporine 0.05% Ophthalmic Emulsion
Number analyzed (Participants) | 36
Scores on a Scale
  Baseline | 1.7 (1.04)
  Change from Baseline at Month 6 (N=32) | -0.8 (1.04)

9. Primary Outcome: Change From Baseline in Reading Rate
Description: Reading speed is assessed as the number of words read correctly in 2 minutes.
Time Frame: Baseline, Month 6
Population: Intent-to-Treat: all enrolled patients who received at least one dose of the study drug
Measure: Mean (Standard Deviation); unit: Words/Minute
Arm/Group | Cyclosporine 0.05% Ophthalmic Emulsion
Number analyzed (Participants) | 40
Words/Minute
  Baseline | 105.2 (17.11)
  Change from Baseline at Month 6 (N=37) | 3.5 (11.69)

10. Primary Outcome: Change From Baseline in Words Read Incorrectly
Description: The numbers of words read incorrectly are counted in 2 minutes. A positive change from baseline indicates a worsening, and a negative change from baseline indicates an improvement.
Time Frame: Baseline, Month 6
Population: Intent-to-Treat: all enrolled patients who received at least one dose of the study drug
Measure: Mean (Standard Deviation); unit: Words
Arm/Group | Cyclosporine 0.05% Ophthalmic Emulsion
Number analyzed (Participants) | 40
Words
  Baseline | 0.4 (0.64)
  Change from Baseline at Month 6 (N=37) | 0.2 (0.90)

11. Primary Outcome: Change From Baseline in Font Size
Description: The minimum font (letter) size read correctly is assessed. Smaller font size indicates better ability. A negative change from baseline indicates an improvement and a positive change from baseline indicates a worsening.
Time Frame: Baseline, Month 6
Population: Intent-to-Treat: all enrolled patients who received at least one dose of the study drug
Measure: Mean (Standard Deviation); unit: Size
Arm/Group | Cyclosporine 0.05% Ophthalmic Emulsion
Number analyzed (Participants) | 40
Size
  Baseline | 12.0 (0.00)
  Change from Baseline at Month 6 (N=37) | -0.2 (0.75)

12. Secondary Outcome: Change From Baseline in OSDI
Description: The OSDI consists of 12 questions measuring the presence of ocular symptoms. Each of the 12 questions is assessed using a 5-point scale (0=none of the time; 4=all of the time). The score is converted to a 0-100 score where 0 is best and 100 is worst. Higher OSDI scores are associated with greater severity. A negative number change from baseline indicates improvement and a positive number change from baseline indicates worsening.
Time Frame: Baseline, Month 6
Population: Intent-to-Treat: all enrolled patients who received at least one dose of the study drug
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Cyclosporine 0.05% Ophthalmic Emulsion
Number analyzed (Participants) | 40
Scores on a Scale
  Baseline | 47.0 (16.97)
  Change from Baseline at Month 6 (N=37) | -19.7 (14.43)

13. Secondary Outcome: Change From Baseline in Ocular Discomfort on a 4-point Scale
Description: Ocular discomfort is assessed on a 4-point scale where 0=no discomfort and 3=most discomfort. A positive number change from baseline indicates a worsening and a negative number change from baseline indicates an improvement.
Time Frame: Baseline, Month 6
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Cyclosporine 0.05% Ophthalmic Emulsion
Number analyzed (Participants) | 40
Scores on a Scale
  Baseline | 2.85 (0.921)
  Change from Baseline at Month 6 (N=37) | -1.30 (1.266)

14. Secondary Outcome: Change From Baseline in Tear Film Break-up Time in the Worse Eye
Description: TFBUT is defined as the time required for dry spots to appear on the surface of the eye after blinking. The longer it takes, the more stable the tear film. A positive number change from baseline indicates improvement and a negative number change from baseline indicates a worsening.
Time Frame: Baseline, Month 6
Population: Intent-to-Treat: all enrolled patients who received at least one dose of the study drug
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Cyclosporine 0.05% Ophthalmic Emulsion
Number analyzed (Participants) | 40
Seconds
  Baseline | 1.55 (0.428)
  Change from Baseline (N=37) | 0.92 (1.044)

15. Secondary Outcome: Change From Baseline in the Interblink Interval in the Worse Eye
Description: The interblink interval measures the time (seconds) between blinks in the worse eye. A positive number change from baseline indicates a worsening (more frequent blinks) and a negative number change from baseline (less frequent blinks) indicates an improvement.
Time Frame: Baseline, Month 6
Population: Intent-to-Treat: all enrolled patients who received at least one dose of the study drug
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Cyclosporine 0.05% Ophthalmic Emulsion
Number analyzed (Participants) | 40
Seconds
  Baseline | 4.18 (3.233)
  Change from Baseline at Month 6 (N=35) | 3.04 (10.637)

16. Secondary Outcome: Change From Baseline in Conjunctival Redness in the Worse Eye
Description: Conjunctival redness is scored in the worse eye on a numeric analog scale ranging from 0=None to 4=Extremely Severe (0.5 increments were allowed). A positive number change from baseline indicates a worsening and a negative number change from baseline indicates an improvement.
Time Frame: Baseline, Month 6
Population: Intent-to-Treat: all enrolled patients who received at least one dose of the study drug
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Cyclosporine 0.05% Ophthalmic Emulsion
Number analyzed (Participants) | 40
Scores on a Scale
  Baseline | 2.06 (0.709)
  Change from Baseline at Month 6 (N=37) | -0.03 (0.707)

ADVERSE EVENTS:
Arm/Group | Cyclosporine 0.05% Ophthalmic Emulsion
Serious Adverse Events (participants affected / at risk) | 2/40
Other Adverse Events (participants affected / at risk) | 12/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cyclosporine 0.05% Ophthalmic Emulsion (N=40)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Renal Failure Acute (Renal and urinary disorders) | 1
Transient Ischaemic Attack (Nervous system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cyclosporine 0.05% Ophthalmic Emulsion (N=40)
Eye Irritation (Eye disorders) | 2
Instillation Site Burn (General disorders) | 3
Instillation Site Pain (General disorders) | 3
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2
Headache (Nervous system disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.